CLINICAL TRIAL: NCT00921323
Title: The Use of Pedometers as an Adjunctive Tool in a School-based Pediatric Weight Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Children's Miracle Network (Other)
Responsible Party: Principal Investigator, Vincent Aluquin, Assistant Professor of Pediatrics, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB Protocol No. 29778
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Obesity
Keywords: Obesity; Physical activity; pedometers; children
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): The control group will be advised to continue to be physically active and record daily steps
  Interventions: Behavioral: Control
- Goal-setting group (Active Comparator): This intervention group would be instructed to increase their daily step count by at least 20% above their baseline gradually over 3 months.
  Interventions: Behavioral: Goal-setting group

INTERVENTIONS:
Behavioral: Goal-setting group — This intervention group will be advised to increase their daily steps by at least 20% gradually over 3 months
  Arms: Goal-setting group
Behavioral: Control — The control group will be advised to continue to be physically active and record daily steps
  Arms: Control

SUMMARY:
The purpose of this study is:

* To validate the use of pedometers in assessing the level of physical activity in middle school children.
* To evaluate whether setting a step goal through the use of pedometers could increase physical activity and prevent weight gain in middle school children.

ELIGIBILITY:
Inclusion Criteria:

* All healthy 8th grade students at the Springboard Academy of the Milton Hershey School willing to participate in the study and whose parents give consent.

Exclusion Criteria:

* Any medical condition that prevents the child from walking during the 12 week study period.
* Non-English speaking student.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Body mass index | 3 months
  BMI will be recorded

SECONDARY OUTCOMES:
Daily step counts | 3 months
  Daily step count will be recorded
Survey questionnaire | 3 months
  Participants will be asked to fill out a survey

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State College of Medicine / Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States